CLINICAL TRIAL: NCT00292487
Title: Isovue and Visipaque in Renally Impaired Patients Undergoing CT
Brief Title: Patients With Renal Impairment Undergoing CT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bracco Diagnostics, Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: IOP107
Record Dates: First submitted 2006-02-14; First posted 2006-02-16 (Estimated); Last update posted 2012-02-08 (Estimated); Status verified 2006-08

CONDITIONS: Contrast Induced Nephropathy

INTERVENTIONS:
Drug: Iopamidol 370 mgI/mL

SUMMARY:
The purpose of the study is to compare the incidence of contrast induced nephrotoxicity following the administration of Isovue or Visipaque in patients with mild to moderate renal impairment who undergo a clinically indicated IV contrast-enhanced (multidetector computed tomography) MDCT of the liver or MDCT angiography of the lower extremities. Serum Creatinine (SCr) will be measured before and up to 48-72 hours post dose.

ELIGIBILITY:
Inclusion Criteria:

* referred for MDCT of liver or peripheral CTA
* stable baseline SCr of 1.5 - 2.5 mg/dL and/or calculated CrCl of 10-60 mL/min

Exclusion Criteria:

* unstable renal function
* required prophylactic drugs to receive contrast (other than hydration)
* uncontrolled diabetes
* currently on dialysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150
Dates: Start 2004-11; Primary Completion 2006-02 (Actual); Study Completion 2006-02 (Actual)

PRIMARY OUTCOMES:
Increase in SCr at 48-72 hours post dose

SECONDARY OUTCOMES:
Compare incidence of delayed hypersensitivity type reactions
Compare changes in heart rate
Compare efficacy of key vessels

CONTACTS AND LOCATIONS:
Overall Officials: Marie Morris, Study Director — Bracco Diagnostics, Inc
Locations (1):
- Bracco Diagnostics, Inc, Princeton, New Jersey, United States